CLINICAL TRIAL: NCT03362190
Title: A Phase 2A Open-label Trial to Assess the Safety of ZIMURA™ (Anti-C5) Administered in Combination With LUCENTIS® 0.5 mg in Treatment Naive Subjects With Neovascular Age Related Macular Degeneration
Brief Title: ZIMURA in Combination With LUCENTIS in Patients With Neovascular Age Related Macular Degeneration (NVAMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH2007
Record Dates: First submitted 2017-10-30; First posted 2017-12-05 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Zimura (previous name); ARC1905; Lucentis; ranibizumab; Wet AMD; avacincaptad pegol; complement factor C5 inhibitor
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Avacincaptad Pegol dosage 1 + Lucentis 0.5 mg
  Interventions: Drug: Avacincaptad Pegol; Drug: Lucentis
- Cohort 2 (Experimental): Avacincaptad Pegol dosage 2 + Lucentis 0.5 mg
  Interventions: Drug: Avacincaptad Pegol; Drug: Lucentis
- Cohort 3 (Experimental): Avacincaptad Pegol dosage 3 + Lucentis 0.5 mg
  Interventions: Drug: Avacincaptad Pegol; Drug: Lucentis
- Cohort 4 (Experimental): Avacincaptad Pegol dosage 4 + Lucentis 0.5 mg
  Interventions: Drug: Avacincaptad Pegol; Drug: Lucentis

INTERVENTIONS:
Drug: Avacincaptad Pegol — Avacincaptad Pegol in combination with Lucentis
  Other Names: Zimura (previous name); IZERVAY; ARC1905
Drug: Lucentis — Avacincaptad Pegol in combination with Lucentis
  Other Names: ranibizumab

SUMMARY:
To assess the safety of intravitreal Zimura™ (complement factor C5 inhibitor) administered in combination with Lucentis® 0.5 mg in treatment naïve subjects with neovascular age related macular degeneration (NVAMD)

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal NVAMD

Exclusion Criteria:

* History or evidence of severe cardiac disease
* Any major surgical procedure within one month of trial entry
* Subjects with a clinically significant laboratory value
* Any treatment with an investigational agent in the past 60 days for any condition
* Women who are pregnant or nursing
* Known serious allergies to the fluorescein dye used in angiography, povidone iodine, to the components of the ranibizumab formulation, or to the components of the Zimura formulation
* Any prior treatment for AMD other than oral supplements of vitamins and minerals

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (23):
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Centers PC, Tucson, Arizona
  - Retina Associates SW, PC, Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Colorado Retina Associates, Golden, Colorado
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Illinois Eye Center, Peoria, Illinois
  - Vitreo Retinal Consultants & Surgeons, Wichita, Kansas
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - VitreoRetinal Surgery, Minneapolis, Minnesota
  - Retina Consultants of Nevada, Henderson, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Retina Vitreous Surgeons of CNY, PC, Syracuse, New York
  - Retina Northwest PC, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Retina Research Institute of Texas, Abilene, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
- Hungary (3):
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Budapest
  - Budapest Retina Associates, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Szemeszeti Klinika, Szeged
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Clinic of Ophthalmology, Riga
  - Dr. Solomatin's eye rehabilitation and vision correction centre, Riga

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26400&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/OPH2007/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Monthly administration of Lucentis 0.5 mg followed 2 days later by Zimura 4mg
- Cohort 2: Monthly administration of Zimura 2mg + Lucentis 0.5 mg administered (given on the same day)
- Cohort 3: Zimura 2mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (Total: 6 doses of Zimura & 3 doses of Lucentis) Maintenance Phase (Month 3-5): Monthly administration of Zimura 2mg + Lucentis 0.5mg given on the same day (Total: 3 doses of Zimura and 3 doses of Lucentis)
- Cohort 4: Zimura 2mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (Total: 6 doses of Zimura & 3 doses Lucentis) Maintenance Phase (Month 3-5): Monthly administration of Zimura 2mg followed 2 days later by Zimura 2mg + Lucentis 0.5mg (Total: 6 doses of Zimura & 3 doses Lucentis)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 10 | 10 | 22 | 22
Completed | 10 | 10 | 22 | 20
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Monthly administration of Zimura 2mg + Lucentis 0.5 mg (given on the same day)
- Cohort 4: Zimura 2mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (6 doses of Zimura and 3 doses of Lucentis) Maintenance Phase (Month 3-5): Monthly administration of Zimura 2mg followed 2 days later by Lucentis 0.5mg + Zimura 2mg (6 doses of Zimura and 3 doses of Lucentis)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 10 | 10 | 22 | 22 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 1 | 5
  >=65 years | 8 | 10 | 20 | 21 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (11.27) | 77.9 (6.62) | 74.1 (7.41) | 78.1 (7.40) | 76.0 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 14 | 12 | 38
  Male | 6 | 2 | 8 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 10 | 21 | 21 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 10 | 22 | 22 | 64
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 0 | 1 | 2 | 3 | 6
  Hungary | 0 | 3 | 8 | 2 | 13
  United States | 10 | 6 | 12 | 17 | 45
ETDRS Visual Acuity -Study Eye [Mean (Standard Deviation); unit: number of letters read] — Visual Acuity reported as the number of letters read on the ETDRS chart by the study eye
  number of letters read | 53.9 (9.0) | 51.5 (5.4) | 52.5 (9.4) | 53.2 (9.9) | 52.8 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Systemic Adverse Events
Description: Number of Participants with systemic treatment-emergent Adverse Events (with calculated percentage)
Time Frame: 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Monthly administration of Zimura 2mg + Lucentis 0.5mg (given on the same day)
- Cohort 4: Zimura 2mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (Total: 6 doses Zimura & 3 doses of Lucentis) Maintenance Phase (Month 3-5): Monthly adminstration of Zimura 2mg followed 2 days later by Zimura 2mg + Lucentis 0.5 mg (Total: 6 doses Zimura & 3 doses of Lucentis)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 22 | 22
Participants
  All causalities | 6 | 5 | 5 | 11
  Related to study drugs | 0 | 0 | 0 | 0

2. Primary Outcome: Ophthalmic Adverse Events
Description: Number of participants with ophthalmic Adverse Events (with calculated percentage)
Time Frame: 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4: Zimura 2mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (Total: 6 doses of Zimura & 3 doses Lucentis) Maintenance Phase (Month 3-5): Monthly administration of Zimura 2mg followed 2 days later by Zimura 2mg + Lucentis 0.5 mg (Total: 6 doses of Zimura & 3 doses Lucentis)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 22 | 22
Participants
  Participants with all causality events in the fellow eye | 1 | 1 | 0 | 2
  Participants with all causality events in the study eye | 8 | 4 | 11 | 15
  Participants with event related to injection procedure in the study eye | 8 | 4 | 10 | 12
  Participants with event related to injection procedure in the fellow eye | 0 | 0 | 0 | 0
  Participants with event related to study drugs in the study eye | 0 | 0 | 0 | 0
  Participants with event related to study drugs in the fellow eye | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Change From Baseline - ECG
Description: Number of patients with a change on their Month 6 ECG when compared to their baseline ECG
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 22 | 22
Participants
  No Change | 7 | 5 | 18 | 12
  Not Clinically Signigicant Change | 3 | 5 | 3 | 6
  Clinically Significant Change | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 1 | 3

4. Other Pre Specified Outcome: Mean Change From Baseline - Study Eye ETDRS Visual Acuity
Description: Mean change from Baseline to Month 6 in the number of letters read by the study eye using the ETDRS Visual Acuity charts. Higher ETDRS letters represents better vision and a larger change in ETDRS letters represents better functioning.
Time Frame: 6 months
Population: safety population
Measure: Mean (Standard Deviation); unit: number of letters read
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 22 | 22
number of letters read | 9.0 (11.0) | 10.2 (18.7) | 10.7 (10.3) | 9.9 (8.2)

5. Other Pre Specified Outcome: Mean Change From Baseline - Vital Signs
Description: Mean change from Baseline to Month 6 in blood pressure (mm Hg). A negative number indicates a decrease and a positive number indicates an increase.
Time Frame: 6 months
Population: safety population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 22 | 22
mm Hg
  Systolic blood pressure (mm Hg) | -12.0 (15.04) | 0.7 (8.92) | -1.9 (14.92) | -5.8 (18.24)
  Diastolic blood pressure (mm Hg) | -3.2 (7.93) | -7.9 (12.32) | -4.7 (11.83) | -0.4 (8.24)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Cohort 1: Monthly administration of Lucentis 0.5 mg followed 2 days later by Zimura 4 mg
- Cohort 2: Monthly administration of Zimura 2 mg + Lucentis 0.5 mg (given on the same day)
- Cohort 4: Zimura 2 mg + Lucentis 0.5 mg Induction Phase (Day 1 - Month 2): Monthly administration of Zimura 2 mg + Lucentis 0.5 mg given on the same day followed 14 days later with Zimura 2mg (Total: 6 doses of Zimura & 3 doses Lucentis) Maintenance Phase (Month 3-5): Monthly administration of Zimura 2mg followed 2 days later by Zimura 2 mg + Lucentis 0.5 mg (Total: 6 doses of Zimura & 3 doses Lucentis)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/22 | 2/22
Other Adverse Events (participants affected / at risk) | 10/10 | 7/10 | 10/22 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=22) | Cohort 4 (N=22)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=22) | Cohort 4 (N=22)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 6 (14) | 1 (1) | 5 (6) | 6 (12)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Punctate keratitis (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (5)
Eye pain (Eye disorders) | 1 (3) | 0 (0) | 0 (0) | 3 (6)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Subretinal fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous opacities (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/PI agrees not to individually publish the results of the Study without IVERIC bio's prior written consent. Institution/PI may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of IVERIC bio.

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03362190/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT03362190/SAP_003.pdf